CLINICAL TRIAL: NCT00996814
Title: Proactive Ethics Intervention to Improve ICU Care
Brief Title: Proactive Ethics Intervention to Improve Intensive Care Unit (ICU) Care
Acronym: PEI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: Principal Investigator, James (Wes) McGaughey, Research Analyst, California Pacific Medical Center Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 26.111EXP
Record Dates: First submitted 2009-09-14; First posted 2009-10-16 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Intensive Care Unit Days
Keywords: Bioethics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proactive Ethics Intervention (Experimental): These patients have an ethics consultant involved in their care beginning on the fifth day of treatment in the ICU
  Interventions: Behavioral: Proactive Ethics Intervention
- Usual Care (No Intervention): These patients receive usual care in the ICU.

INTERVENTIONS:
Behavioral: Proactive Ethics Intervention — The ethicist will: 1) meet with the patient or surrogate to assess the case and the decision-making capacity of the patient; 2) make an ethical diagnosis, framing the issues in easily understood ethical terms with the involved parties; 3) recommend the next steps, including measures to improve communication. The ethicist will help to articulate consensus or disagreement and either facilitate implementing the consensus or facilitate ways to address and resolve disagreements; 4) document the consultation in the patient's medical record, identifying the ethical issues identified, the steps taken to address those issues, the options and ethical rationales considered, the outcome and the future plan; 5) follow-up to provide ongoing support and record a follow up progress note in the chart; and 6) participate in evaluation.
  Arms: Proactive Ethics Intervention

SUMMARY:
The primary aim of the study is to demonstrate the value of a preemptive approach to ethics consultation in an ICU. The investigators hope to answer the question: Will proactive ethics interventions by a skilled and experienced ethicist, participating in treatment discussions with physicians and nurses, as well as discussions with patients/surrogates, improve the quality of ICU care experienced by patients requiring prolonged treatment in the ICU (5 days or longer) by increasing their perceived quality of care and reducing the length of stay in the ICU by non-survivors?

The study is a randomized trial of the use of an ethics consultant to address latent or manifest ethical issues in patients who remain in the ICU for five days or more, as compared to usual care. The investigators are testing the hypothesis that expanding the role of ethics consultations in the ICU to make them proactive will improve the process and outcomes of patient care by shortening the length of stay in non-survivors, and reducing suffering and unwanted and/or unnecessary aggressive treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adult (over 18 years of age)
* Under treatment for five days or more in the ICU

Exclusion Criteria:

* Under the age of 18
* Non-English Speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2007-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Length of Stay in Days | Date and time of admission to date and time of discharge (in 24 hour periods)

SECONDARY OUTCOMES:
Patient Satisfaction | Survey administered every two days while patient is in the ICU and a final survey one month after discharge from the hospital
Provider satisfaction | Survey administered daily while patient in under their care and 48 hours after their patient's discharge

CONTACTS AND LOCATIONS:
Overall Officials: William S Andereck, MD, Principal Investigator — California Pacific Medical Center; Lawrence J Schneiderman, MD, Principal Investigator — University of California, San Diego; J. Westly McGaughey, B.A., Principal Investigator — California Pacific Medical Center; Albert R. Jonsen, Ph.D., Principal Investigator — California Pacific Medical Center
Locations (1):
- California Pacific Medical Center, San Francisco, California, United States

REFERENCES:
- [Derived] Andereck WS, McGaughey JW, Schneiderman LJ, Jonsen AR. Seeking to reduce nonbeneficial treatment in the ICU: an exploratory trial of proactive ethics intervention*. Crit Care Med. 2014 Apr;42(4):824-30. doi: 10.1097/CCM.0000000000000034. PMID 24201177